CLINICAL TRIAL: NCT05322356
Title: Interstitial Brachytherapy of the Prostate With Iodine 125 Implant With Target Dose Supplementation in the Tumor Volume Guided by the TRINITY® PERINE 3D Ultrasound System
Brief Title: Prostate Interstitial Brachytherapy With I125 Implant With Target Dose Supplementation in the Tumor Volume Guided by TRINITY® PERINE 3D System
Acronym: FOCUS-BOOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Koelis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-A01178-33
Record Dates: First submitted 2021-11-24; First posted 2022-04-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
Keywords: Interstitial brachytherapy; Iodine 125 implant; 3D TRINITY® Perine system
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Iodine-125

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Interstitial Brachytherapy of the Prostate With Iodine 125 Implant With Target Dose Supplementation in the Tumor Volume Guided by the TRINITY® PERINE 3D system
  Interventions: Other: Interstitial Brachytherapy of the Prostate With Iodine 125 Implant With Target Dose Supplementation in the Tumor Volume Guided by the TRINITY® PERINE 3D

INTERVENTIONS:
Other: Interstitial Brachytherapy of the Prostate With Iodine 125 Implant With Target Dose Supplementation in the Tumor Volume Guided by the TRINITY® PERINE 3D — Target dose supplement with the TRINITY® PERINE 3D system

SUMMARY:
The objective of the FOCUS-Boost project is to implant for the first time with a 3D ultrasound image fusion registration system (3D echo) implant of iodine 125 with precision in a target volume determined by positive biopsies.

DETAILED DESCRIPTION:
The interstitial brachytherapy procedure for the prostate does not allow for a robust focal treatment to accurately deliver additional dose to the tumour volume. FOCUS BOOST allows the precise implantation of 125 iodine implant with greater accuracy (using a 3D ultrasound image fusion registration system) in a target volume.

For this purpose, positive biopsies, performed in this research protocol, will be used prior to surgery. Prostate brachytherapy will be optimised thanks to the TRINITY® system and its guidance quality, by increasing the dose of the intra-prostate tumour volume (BOOST) without increasing the total dose delivered to the prostate. Increasing the dose to the tumour target volume could improve disease control and decrease the risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Patient to be treated with brachytherapy
* Patient with low or favorable intermediate risk prostate adenocarcinoma ISUP 1 and 2, G6 (3+3) or G7 (3+4)
* Life expectancy of more than 10 years
* PSA (prostate-specific antigen) < 15 ng/ml
* cT1c or cT2a or cT2b
* Prostate volume ≤ 60 cc
* ECOG Performance status 0-2
* Patient is affiliated to a health insurance system
* Patient who has signed consent form

Exclusion Criteria:

* Patient with urinary function disorders IPSS> 14
* Prostate volume > 60cc.
* Gleason 7(4+3) or Gleason score ≥8
* PSA ≥ 15 ng/ml
* Patient with metastases
* Hormone therapy with antiandrogen or LHRH analogue
* History of abdominopelvic irradiation
* Inflammatory digestive disease (haemorrhagic rectocolitis, Crohn's disease)
* Interventional study in progress that may interfere with the present study
* Protected persons (patient concerned by articles L1121-5, L1121-6, L1121-8 of the French public health code)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Implant for the first time, in a clinical situation, iodine 125 implants in a planned target volume, using a 3D echo-mapping fusion guidance system of positive biopsies. | 24 hours
  To evaluate the number of successful/failed iodine 125 implants (BOOST implants) implanted in the CTV-boost (Clinical Target Volume) defined from the mapping of positive biopsies.
  The maximum number of BOOST implant implanted will be 4 implants, depending on the size of the target:
  10 mm< target ≤ 15 mm = 2 implants; 15 mm < target ≤ 20mm = 3 implants; 20 mm < target ≤ 30 mm = 4 implants; Success is defined as "the centre of the implant is in the target volume". Failure is defined as "the centre of the implant is outside the target volume". The primary endpoint is evaluated on the ultrasound acquisition performed with the Trinity® Perine probe, at the end of the BOOST implant insertion procedure

SECONDARY OUTCOMES:
Assess toxicity (pre brachytherapy visit, M1, M3, M6, M12), with questionnaires | 12 months
  Assessment of toxicity by questionnaires (IPSS score + urinary symptom quality of life).
  IPSS:: International Prostate Score Symptom (0 to 35: Score 20-35: severely symptomatic. Score 8-19: moderately symptomatic)
Assess toxicity (pre brachytherapy visit, M1, M12) with flowmetry | 12 months
  Assessment of toxicity by urinary flowmetry
Assess toxicity (pre brachytherapy visit, M1, M3, M6, M12) with CTCAE score | 12 months
  Assessment of toxicity by classification of toxicities according to CTCAE score (Common Terminology Criteria for Adverse Events: Grade 1 Mild / Grade 2 Moderate / Grade 3 Severe or medically significant but not immediately life-threatening / Grade 4 Life-threatening consequences / Grade 5 Death related to A
To assess the efficacy of the treatment at M6 and M12. | 12 months
  PSA (Prostate Specific Antigen) test
To check the absence of overdose in the prostate at D0 and M1. | 1 month
  V150% < 60% of prostate volume on CT dosimetry at D0 and 1 month
To check the absence of overdose in organs at risk (bladder, urethra, rectum) at D0 and M1. | 1 month
  Absence of overdose in organs at risk on scanner dosimetry
Dose to CTV-dosi at 150% | 1 month
  V150% > 95% for CTV-dosi (on Variseed dosimetry) at J0
Assess quality of life (inclusion, M1, M3, M6, M12). | 12 months
  QLQ-C30 (Quality of Life Questionnaire) score
Assess sexual health (inclusion, M1, M3, M6, M12). | 12 months
  IIEF5 questionnaire score (Erectile dysfunction severe (score 5-10), moderate (11-15), mild (16-20), normal erectile function (21-25) and uninterpretable (1-4)).
Measure the duration of the complete procedure, the additional act (BOOST) and the final ultrasound acquisition performed at the end of the procedure (when performed). | 24 hours
  Duration of the entire procedure, the additional procedure (BOOST), and the final ultrasound acquisition at the end of the procedure (when performed)
(For the last 5 patients): Estimate the quality of the registration after insertion of the implants. | 24 hours
  (For the last 5 patients): Final ultrasound acquisition performed at the end of the procedure with the Trinity® Perine system

CONTACTS AND LOCATIONS:
Overall Officials: Carole Iriard, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Isabelle Boudry, Grenoble, France

REFERENCES:
- See also: Centre d'Investigation Clinique Innovation Technologique — https://www.cic-it.fr/cic-it-grenoble.php